CLINICAL TRIAL: NCT00527072
Title: A Multicenter, Open-label Study to Assess the Efficacy and Safety of Infliximab (REMICADE�) Therapy in Patients With Plaque Psoriasis Who Had an Inadequate Response to Etanercept (ENBREL�)
Brief Title: PSUNRISE - Prospective Study Using Remicade in Psoriasis Patients With an Inadequate Response to Etanercept
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centocor Ortho Biotech Services, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR014500; C0168Z04 (Other: Centocor Ortho Biotech Services, L.L.C.)
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Results first posted 2010-06-24 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Psoriasis
Keywords: plaque psoriasis; psoriasis; infliximab; remicade; etanercept; enbrel; psunrise; C0168Z04
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): infliximabOpen-label 5 mg/kg infliximab infusions at Weeks 0, 2, 6, 14, and 22.
  Interventions: Biological: infliximab

INTERVENTIONS:
Biological: infliximab — Open-label 5 mg/kg infliximab infusions at Weeks 0, 2, 6, 14, and 22.

SUMMARY:
The purpose of this study is to test the safety and effectiveness of infliximab in patients with plaque psoriasis who have been receiving the drug etanercept for treatment of their plaque psoriasis for at least four months, without enough improvement in their psoriasis symptoms.

DETAILED DESCRIPTION:
The most common form of psoriasis is plaque-type psoriasis, which is characterized by recurrent flaring of thickened, red, scaly patches of skin. Although psoriasis is usually not life threatening, these physical discomforts combined with the potential psychological effects of the disease may interfere with everyday activities and negatively impact an individual's quality of life. Many therapies are available for psoriasis; however, with limited effectiveness and significant toxicity. Infliximab is an antibody made in a laboratory. Antibodies are proteins that fight other substances in the body that may cause infections or diseases. A substance called "tumor necrosis factor" (TNF) naturally occurs in the body. TNF is related to the itchy patches of skin (or plaques) of psoriasis. Infliximab stops the TNF from working. Other studies have shown that stopping the TNF may reduce the plaques. To address the unmet medical need for effective chronic therapies, TNFalpha blockers have recently been used to treat patients with moderate to severe plaque psoriasis. Etanercept also works by stopping the TNF, but in a different way than infliximab. This multi-center, open-label study is designed to test whether or not patients with plaque psoriasis who have not responded well to etanercept treatment may benefit from treatment with infliximab. Key effectiveness measurements will include the time to onset of symptom improvement and health-related quality of life. Safety will be assessed throughout the study. Two weeks after their last dose of etanercept, all eligible patients will receive open-label 5 mg/kg infliximab infusions at Weeks 0, 2, 6, 14, and 22.

ELIGIBILITY:
Inclusion Criteria:

* Have plaque psoriasis despite at least 4 months of treatment with etanercept per current product labeling
* Have psoriatic target lesions that have a PGA score greater than 1 (minimal) at screening
* If receiving methotrexate at screening, must have received methotrexate for at least 3 months and at a stable dose of <= 25 mg/week for at least 4 weeks prior to screening
* If receiving cyclosporine at screening, must have received cyclosporine at a stable dose of <= 5 mg/kg daily for at least 4 weeks prior to screening.

Exclusion Criteria:

* Have already received infliximab or adalimumab
* Have shown a previous immediate hypersensitivity response, including anaphylaxis, to an immunoglobulin product
* Have a history of latent or active granulomatous infection, including tuberculosis, histoplasmosis, or coccidioidomycosis, prior to screening
* Have a concomitant diagnosis or any history of Congestive Heart Failure
* Are pregnant, nursing, or planning pregnancy
* Have used systemic corticosteroids within the 4 weeks prior to screening
* Have used topical corticosteroids or have initiated treatment with other topical therapies that could affect psoriasis or Psoriasis Area and Severity Index (PASI) evaluation (e.g., tar, anthralin, calcipotriene, tazarotene, methoxsalen) within 2 weeks prior to screening
* Have used new systemic agents/treatments, other than methotrexate, that can affect psoriasis including, but not limited to, immunosuppressants and/or psoralen plus ultraviolet A light (PUVA) within the 4 weeks prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Centocor Ortho Biotech Services, L.L.C. Clinical Trial, Study Director — Centocor Ortho Biotech Services, L.L.C.

REFERENCES:
- [Derived] Gottlieb AB, Kalb RE, Blauvelt A, Heffernan MP, Sofen HL, Ferris LK, Kerdel FA, Calabro S, Wang J, Kerkmann U, Chevrier M. The efficacy and safety of infliximab in patients with plaque psoriasis who had an inadequate response to etanercept: results of a prospective, multicenter, open-label study. J Am Acad Dermatol. 2012 Oct;67(4):642-50. doi: 10.1016/j.jaad.2011.10.020. Epub 2011 Dec 9. PMID 22153792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 217 subjects enrolled into the study but 2 subjects did not receive any study medication so they were excluded from analysis.
Period: Overall Study
Arm/Group | Infliximab
Started | 215
Completed | 179
Not Completed | 36
Not completed — Adverse Event | 13
Not completed — Lack of Efficacy | 11
Not completed — Lost to Follow-up | 3
Not completed — Protocol Violation | 2
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 198
  >=65 years | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 44.4 (13.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 137

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve a Physician Global Assessment (PGA) Score of Minimal (1) or Clear (0)
Description: Patients who did not have a PGA score at Week 10 will be treated as not having achieved a PGA score of minimal (1) or clear (0) at Week 10. Specifically, treatment failures prior to Week 10 will be classified as not having a minimal (1) or clear (0).
Time Frame: Week 10
Population: This analysis is based on the evaluable population that includes the all enrolled patients who received at least one infliximab infusion, and had a baseline PGA score greater than 1.
Measure: Number; unit: participants
Groups:
- Infliximab: Open-label study, patients received IV infusions of 5 mg/kg infliximab at Weeks 0, 2, 6, 14, and 22
Arm/Group | Infliximab
Number analyzed (Participants) | 211
participants | 138 [58.6 to 71.8]
Statistical Analysis 1: Comparison: Infliximab; null hypothesis H0: proportion = 0.30; Test type: Superiority or Other; p = 0.05, exact binomial distribution; Proportion = 0.654, 95% CI 2-sided [0.586 to 0.718]

2. Secondary Outcome: Number of Patients Achieved Psoriasis Area Activity Index (PASI) 50 Response at Week 10
Description: A PASI 50 responder is defined as a patient who has achieved at least a 50% improvement in the overall PASI score from baseline. PASI is an index used for assessing and grading the severity of psoriatic lesions and their response to therapy. The PASI produces a numeric score that can range from 0 to 72. A score less than 10 signifies a mixture of mild and moderate disease; a score greater than 10 but less than or equal to 30 signifies moderate disease; and a score greater than 30 signifies severe disease.
Time Frame: Week 10
Population: Analysis is based on observed mITT (modified Intent to Treat) patients. Treatment failures are classified as not achieving a PASI 50, 75, 90, or 100 response at all visits after the date of treatment failure. For non-treatment failure patients who did not have a PASI score at the visit due to other reasons, will not have data imputed at that visit.
Measure: Number; unit: participants
Arm/Group | Infliximab
Number analyzed (Participants) | 211
participants | 167 [73.0 to 84.4]
Statistical Analysis 1: Comparison: Infliximab; Test type: Superiority or Other; p = 0.05, exact binomial distribution; proportion = 0.791, 95% CI 2-sided [0.730 to 0.844]

3. Secondary Outcome: Number of Patients Achieved Psoriasis Area Activity Index (PASI) 50 Response at Week 26
Time Frame: Week 26
Population: This analysis is based on all observed mITT patients. The treatment failures will be classified as not achieving a PASI 50, 75, 90, or 100 response at all visits after the date of treatment failure. For non-treatment failure patients who did not have a PASI score at the visit due to other reasons, their data at that visit will not be imputed.
Measure: Number; unit: participants
Arm/Group | Infliximab
Number analyzed (Participants) | 209
participants | 135 [57.7 to 71.1]
Statistical Analysis 1: Comparison: Infliximab; Test type: Superiority or Other; p = 0.05, exact binomial distribution; proportion = 0.646, 95% CI 2-sided [0.577 to 0.711]

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of patient informed consent until the Week 30 follow-up assement, for each patient.
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 8/215
Other Adverse Events (participants affected / at risk) | 63/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=215)
Myocardial ischaemia (Cardiac disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Bursitis infective (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Convulsion (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infliximab (N=215)
Upper respiratory tract infection (Infections and infestations) | 21
Nasopharyngitis (Infections and infestations) | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 19
Headache (Nervous system disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days